CLINICAL TRIAL: NCT00849303
Title: Gait-Oriented Rehabilitation at Different Phases in Patients With Acute Stroke - Multicenter Randomized Controlled Trial.
Brief Title: Multicenter Rehabilitation Study in Acute Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jyvaskyla (Other)
Collaborators: Northern Savo Hospital District (Other); Academy of Finland (Other); Brain Research and Rehabilitation Center Neuron (grant # 1/2009) (Unknown)
Responsible Party: Sinikka H Peurala, Post doctoral researcher, University of Jyväskylä/Department of Health Sciences/Finnish Centre for Interdisciplinary Gerontology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5772765; Academy of Finland 114291
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; gait; timing; transcranial magnetic stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- earlier gait-oriented rehabilitation (Experimental): Patients practise walking every workday for 60 min (actual 30min) either on a treadmill or on a gait trainer for four weeks, and receive also other physiotherapy 60 min daily.
  Interventions: Other: gait-oriented rehabilitation
- later gait-oriented rehabilitation (Active Comparator): Patients practise walking every workday for 60 min (actual 30min) either on a treadmill or on a gait trainer for four weeks, and receive also other physiotherapy 60 min daily.
  Interventions: Other: gait-oriented rehabilitation

INTERVENTIONS:
Other: gait-oriented rehabilitation — Patients practise walking every workday for 60 min (actual 30min) either on a treadmill or on a gait trainer for four weeks, and receive also other physiotherapy 60 min daily.Patients starts within 10 days since stroke onset.
  Arms: earlier gait-oriented rehabilitation
Other: gait-oriented rehabilitation — Patients practise walking every workday for 60 min (actual 30min) either on a treadmill or on a gait trainer for four weeks, and receive also other physiotherapy 60 min daily.Patients starts five weeks after stroke onset.
  Arms: later gait-oriented rehabilitation

SUMMARY:
The purpose of the first part of this study is to understand plastic brain mechanisms associated with successful gait-oriented stroke rehabilitation. Patients are randomized to receive intensive in-patient multiprofessional rehabilitation at different time points. One group will receive rehabilitation immediately after an acute care at the neurological clinic (8 days) and one group 5 weeks after the insult. Patients practise walking every workday for 60 min (actual 30min) either on a treadmill or on a gait trainer for four weeks, and receive also other physiotherapy. In addition to selected parameters measuring brain plasticity, detailed assessments of functional abilities including motor ability and quality of life will be performed. A novel tool, MR-image navigated transcranial magnetic stimulation (TMS) is utilized in assessing cortical excitability in relation to stroke, time, rehabilitation, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* first supratentorial stroke or no significant disturbance from an earlier stroke (Modified Ranking Scale, MRS 0-2)
* time since onset of stroke no more than 10 days
* Functional Ambulatory Category (FAC) 0-3
* voluntary movement in the leg of the affected side
* Barthel Index (BI) 25-75 points- no unstable cardiovascular disease
* Body Mass Index (BMI) <32
* no severe malposition of joints
* no severe cognitive or communicative disorders
* no other health-related or social barriers to participate intensive rehabilitation

Exclusion Criteria:

* ICH, or MRS >2
* time since onset of stroke more than 10 days
* FAC >3
* no voluntary movement in the leg of the affected side
* BI <25 or >75
* severe malposition of joints
* severe cognitive or communicative disorders

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulatory Category | 4 measures during six months
Barthel Index | 4 measures during 6 months

SECONDARY OUTCOMES:
10 meters's walking speed | 4 measures during 6 months
6 minutes' walking distance | 4 measures during 6 months
Berg Balance Scale | 4 measures during 6 months
Functional Status Questionnaire | 4 measures during 6 months
Geriatric Depression Scale -15 | 4 measures during 6 months
Beck Depression Intervention modified by Raitasalo | 4 measures during 6 months
Modified Motor Assessment Scale | 4 measures during 6 months
Postural sway by Good Balance | 3-4 measures during 6 months
spatio-temporal gait analysis by GaitRite | 3-4 measures during 6 months
WHOQOF-BREF | at end and at 6 months' follow-up
TMS responses (MT,MEPs,SP,SICI) | 4 measures during 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Middle Finland central hospital and Kinkomaa hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Brain Research and Rehabilitation Center Neuron, Kuopio
  - Tampere university hospital, Tampere